CLINICAL TRIAL: NCT03166072
Title: Health Education vs Meditation in Irreversible Age-Related Vision Loss Patients and Their Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 111334
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Low Vision, One Eye, Unspecified Eye; Low Vision Blindness
Keywords: Irreversible age-related vision loss; Randomized controlled trial; Meditation; Pilot study; Quality of life
MeSH Terms: conditions — Vision, Low | interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meditation (Active Comparator): Participants randomized to this arm will undergo the MEDITATION intervention, with weekly training and reinforcement sessions.
  Interventions: Other: Meditation
- Treatment as Usual (No Intervention): Participants randomized to this arm will continue to undergo the usual standard of care. The usual standard of care for IARVL patients includes no active treatment since eye surgeons have done all that could possibly be done to restore vision.
- Health Enhancement Program (HEP) (Other): Participants randomized to this arm will undergo the Health Enhancement Program (HEP) intervention, with weekly sessions identical in structure to those of the MEDITATION arm.
  Interventions: Other: Health Enhancement Program

INTERVENTIONS:
Other: Meditation — This therapy will be delivered using the hospital approved Microsoft TEAMS platform by trained, certified non-clinician teachers. 25 irreversible age-related vision loss patients and their 25 caregivers in the MEDITATION arm will be trained for 2 consecutive days (2 hours/day) in the first week, followed by 1-hour weekly reinforcement sessions for 11 weeks. Participants will learn how to respond to experiences that arise in meditation, will discuss what enhances or detracts from effective meditation, and review methods for meditating at home. Weekly reinforcement sessions will include 33 minutes of guided meditation practice, and then focus on participants' experiences with meditation during the week, additional observations, and a review of relevant knowledge to support their home practice. Each of these follow-up sessions will include a 33-minute guided meditation session. Participants will also be encouraged to practice daily at home for 33 minutes per session.
  Arms: Meditation
Other: Health Enhancement Program — HEP was designed and used as a manualized active control in meditation-based intervention trials. We have tailored HEP to be structurally equivalent to MEDITATION intervention, with similar-sized groups, meeting for 2 days for 2 hours, and then one 60-75-minute follow up session weekly for the subsequent 11 follow ups. Participants allocated to HEP will be completing the same amount of home practice as MEDITATION, and will be asked to complete weekly practice logs. Participants will learn about health promotion, including the benefits of a lifestyle of healthy diet, music, recreation, and exercise, but will not learn breathing techniques, or meditation. In HEP, which is provided according to specific guidelines for administration, participants get the support of a group and facilitator, and talk through and try to implement positive health-enhancing life changes.
  Arms: Health Enhancement Program (HEP)

SUMMARY:
Investigators aim to assess the feasibility of delivering two augmentation interventions, Meditation and a Health Enhancement Program, for potentially enhancing the quality of life and mental health of Irreversible Age-Related Vision Loss (IARVL) patients and/or their caregivers.

DETAILED DESCRIPTION:
Using a mixed-method design, a pilot randomized controlled trial (RCT) study, investigators aim to assess the feasibility of delivering two augmentation interventions, Meditation to Remove Stress and Create Proper System in Mind (MEDITATION) and a Health Enhancement Program (HEP) for potentially enhancing the quality of life and mental health of Irreversible Age-Related Vision Loss (IARVL) patients and/or their caregivers. MEDITATION is a standardized, manualized therapy where participants will be guided by an instructor on meditation techniques, followed by weekly reinforcement sessions. HEP is a similarly structured intervention that controls for several factors experienced in the MEDITATION group, such as group support and morale, behavioral activation, reduction of stigma, facilitator attention, treatment duration, and time spent on at-home practice. Participants will learn about health promotion, including the benefits of a lifestyle of healthy diet, music, recreation, and exercise, but will not learn breathing techniques, or meditation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with irreversible age-related vision loss (IARVL) and have ongoing significant disability and/or their caregivers who agree to consent.
* IARVL patients between age 60 to 85 years or caregivers between 18 to 85 years.
* Deemed competent to provide individual consent to participate.
* Speak and understand English without requirement for interpretation or assistance.
* Have no significant self-reported or physician diagnosed mental health disorder other than depressive and/or anxiety symptoms.
* Have either a minimum of CES-D 20-item scale score of 16 OR a minimum of 8 on the Hospital Anxiety Scale (HADS-A) 7-item sub-scale.
* Have sufficient hearing to be able to follow verbal instructions
* Ability to sit independently without physical discomfort for 30 minutes.
* Willing and able to attend, via Microsoft TEAMS software, the four initial training sessions of MEDITATION or HEP and at least 6 follow-up sessions.
* Willing to dedicate 33 minutes per day to their assigned home practice.

Exclusion Criteria:

* Inability to provide informed consent.
* Dementia as defined by MoCA < 21.
* Have significant suicidal ideation as per self-report (CES-D = 3 on item question 14 and/or 15).
* Have severe depression CES-D ≥ 24.
* Participating in other similar studies.
* Have a lifetime diagnosis of self-reported other mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
* Self-reported substance abuse or dependence within the past 3 months.
* Have an acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.
* Have a terminal medical diagnosis with prognosis of less than 12 months.
* Having any planned changes to mood-altering medications at the time of enrollment for the next 12 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-04-20 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Participants screened | Through study completion, an average of 1 year
  Number of participants screened
Participants enrolled | Through study completion, an average of 1 year
  Proportion of patients and caregivers who enrol in the study after screening
Retention rate | Up to 12 weeks.
  Rate of participation retention in the study
Adherence rate | Up to 12 weeks
  Rate of adherence to study protocol
Assessment rating and duration | Up to 12 weeks
  Proportion of planned ratings that are completed and duration of assessment visits
Intervention cost | Up to 12 weeks
  Intervention cost per case
Data quality | Up to 12 weeks
  Completeness and quality of final data for analysis

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQOL) | Up to 12 weeks
  Improvement in HRQOL score as measured by the Short Form 12 Health Survey (SF-12) up to 12 weeks.
Number of participants approached | Through study completion, an average of 1 year
  Number of potential participants (IARVL patients and their caregivers) approached per month
Change in vision-related quality of life (VRQOL) | Up to 12 weeks
  Improvement in VRQOL score as measured by the Visual Function 14-item questionnaire (VF-14) up to 12 weeks.
Change in depression score | Up to 12 weeks
  Reduction in depressive symptoms as measured by the Center for Epidemiological Studies Depression questionnaire (CES-D) scores up to 12 weeks.
Change in anxiety score | Up to 12 weeks
  Reduction in anxiety symptoms as measured by the Hospital Anxiety Scale questionnaire (HADS-A) scores up to 12 weeks.
Change in sleep quality | Up to 12 weeks
  Enhanced sleep quality as measured by reduction in Pittsburg Sleep Quality Index questionnaire (PSQI) scores (≤ 5) up to 12 weeks.
Change in community integration | Up to 12 weeks
  Enhanced community integration as measured by an increase in Community Integration Questionnaire (CIQ) scores up to 12 weeks.
Change in caregiver burden | Up to 12 weeks
  Reduced caregiver burden as measured by reduction in Zarit Burden Interview (ZBI) scores up to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers since the current research team has the necessary expertise to conduct data analysis.